CLINICAL TRIAL: NCT03374943
Title: A Phase I Safety and Bioimaging Trial of KB004 in Patients With Glioblastoma
Brief Title: A Trial of KB004 in Patients With Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2017-002
Record Dates: First submitted 2017-09-26; First posted 2017-12-15 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — KB004

STUDY DESIGN:
Intervention Model Description: The study will use a 3+3 methodology for the 3 dose levels proposed. In brief, three patients will be recruited per dose level. In the absence of any Dose Limiting toxicity (DLT) in a cohort, escalation to the next dose level will occur.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KB004 dose escalation (Experimental): Patients will be entered at each KB004 dose level sequentially until 3-6 patients are evaluable for safety. Three sequential cohorts are planned in this study (3.5mg/kg, 5.25 mg/kg, 7.9 mg/kg) Additional dose levels may be explored based on the emerging data in the study.
  Interventions: Drug: KB004

INTERVENTIONS:
Drug: KB004 — KB004 is a recombinant, non-fucosylated, IgG1κ (human f-allotype) monoclonal antibody targeting the extracellular ligand binding domain of the EphA3 (ephrin receptor) tyrosine kinase

SUMMARY:
This is a study of drug KB004 in patients with recurrent glioblastoma (GBM). Eligible patients with measurable tumours will receive an initial trace (5mg) dose of zirconium labelled KB004 (89ZrKB004) on day 1 followed by sequential Positron emission tomography (PET) imaging over 1 week to determine its biodistribution into GBM and normal tissues. Safety assessments and pharmacokinetic (movement of drug) sampling will also be undertaken over this time. On Day 8, patients commence weekly KB004 infusions over 2 hours with standard premedications. Three cohorts are planned in this study (3.5mg/kg, 5.25 mg/kg, 7.9 mg/kg; additional dose levels may be explored based on toxicity, efficacy and biodistribution data as determined by the safety monitoring committee). On day 36, patients receive both 89ZrKB004 and KB004, allowing assessment of receptor occupancy to guide recommended phase two dose (RPTD) determination. Response rate (RANO) and survival data will be collected and patients benefiting may continue KB004 treatment until disease progression. Primary objective: to determine the toxicity and recommended phase two dose (RPTD) of KB004 in patients with advanced Glioblastoma (GBM).

Secondary objectives: to determine the biodistribution and pharmacokinetics of 89ZrKB004; to determine frequency of EphA3 (ephrin receptor A3) positive glioblastoma in archival specimens and by 89ZrKB004 scans, and correlate with known biomarkers; to describe response rates per RANO criteria (Response Assessment in Neuro-Oncology Criteria) and pharmacodynamics following KB004 infusion; Exploratory objectives: to perform exploratory analysis between clinical outcomes and biodistribution/Pharmacokinetics (PK)/pharmacodynamics (PD) data, including from matched biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (greater than or equal to 18 years of age) with histologically proven glioblastoma
* Evidence of progressive glioblastoma (if within 3 months of radiotherapy, then progression outside of radiotherapy field is required)
* Measurable disease by RANO (Response Assessment in Neuro-Oncology Criteria)
* ECOG (Eastern Cooperative Oncology Group score) 0 to 1
* Expected survival more than 3 months
* Steroid dose less than 2.5 mg per day dexamethasone equivalents and stable or reducing for 1 week prior to day 1
* Archived (formalin fixed paraffin embedded) tissue or frozen tumour tissue or consent to obtain a fresh tumour biopsy at enrolment is required.
* Adequate organ function. Out of range values that are not clinically significant will be permitted, except for the following laboratory parameters which must be within the ranges specified
* Neutrophils greater than or equal to 1.5 x 109 per L
* Platelets greater than or equal to 100 x 109 per L
* International Normalised Ratio less than or equal to 1.4
* Serum Aspartate aminotransferase and Alanine aminotransferase less than or equal to 2.5 x ULN (upper limit of normal)
* Serum bilirubin less than or equal to 1.5 x ULN (upper limit of normal)

Exclusion Criteria:

* Evidence of infratentorial, extracranial or leptomeningeal disease
* More than one prior systemic therapy for progressive disease or prior Steriotactic radiosurgery (SRS) to sites of GB (glioblastoma).
* Prior treatment with bevacizumab or gliadel wafers
* Evidence of current or prior intracranial hemorrhage
* Need for anti-platelet or anti-coagulant drugs
* Use of anti-cancer therapy including craniotomy, chemotherapy, immunotherapy, radiotherapy, or any investigational therapy within 28 days prior to Study Day 1
* History of major immunologic reaction to any immunoglobulin G containing agent
* Medical conditions which place the subject at an unacceptably high risk
* Subject is pregnant, lactating or unwilling or unable to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With KB004 Treatment-Related Adverse Events as Assessed using CTCAE v4.0. To determine the maximum tolerated dose (MTD). | 0-24 months
  Three patients are recruited per dose level, 3 dose levels. Dose limiting toxicity (DLT) defined as Grade 4 neutropenia > 7 day duration Grade 3 or 4 febrile neutropenia Grade 3 or 4 thrombocytopenia > 7 day duration Grade 4 anaemia > 7 day duration Grade 3 or 4 non-hematologic adverse events which do not resolve within 48 hours with maximal supportive care.
  Grade 4 or recurrent Grade 3 infusion reactions despite maximal supportive care and dose reductions Significant intracranial haemorrhage not reasonably attributed to other cause More than 14 days of treatment delay due to attributable toxicity Other toxicities as determined by the investigators. In the absence of any dose limiting toxicity in a cohort, escalate to the next dose level. If one DLT is seen in the first three patients of a cohort, an additional three patients will be recruited to that cohort. If two or more DLT's are seen in any cohort, that cohort will be deemed the maximum tolerated dose.

SECONDARY OUTCOMES:
Biodistribution of 89Zr-KB004 | 0-24 months
  Eligible patients with measurable tumours will receive an initial trace (5mg) dose of zirconium labelled KB004 (89Zr-KB004) on day 1 followed by sequential Positron emission tomography, or PET imaging over 1 week to determine its biodistribution into GBM and normal tissues, frequency of EphA3 (ephrin type-A receptor 3) expression in glioblastoma (GBM) and quantitative tumor antibody uptake.
Response rates following KB004 infusion | 0-24 months
  Response Assessment in Neuro-Oncology criteria will be used to interpret MRI (magnetic resonance imaging) scans
Plasma concentration versus time (Serum half life) of 89Zr-KB004 | 0-43 days
  Pharmacokinetics (plasma concentration versus time) of 89Zr-KB004 will be determined using gamma well counting of the Zirconium in the samples at various timepoints-Day 1 89Zr-KB004 infusion: pre-infusion, 5min, 1 hour, 2 hours, 4 hours and 24 hours post infusion, then Day 3 or 4, 6 or 7. PK (Pharmacokinetics) timepoints Day 89Zr-KB004 infusion: pre-infusion, 5min, 1 hour, 2 hours, 4 hours and 24 hours post infusion then Day 39 or 40 and Day 42 or 43.
Cmax of 89Zr-KB004 | 0-43 days
  Pharmacokinetics (Cmax) of 89Zr-KB004 will be determined using gamma well counting of the Zirconium in the samples at various timepoints-Day 1 89Zr-KB004 infusion: pre-infusion, 5min, 1 hour, 2 hours, 4 hours and 24 hours post infusion, then Day 3 or 4, 6 or 7. PK (Pharmacokinetics) timepoints Day 89Zr-KB004 infusion: pre-infusion, 5min, 1 hour, 2 hours, 4 hours and 24 hours post infusion then Day 39 or 40 and Day 42 or 43.

OTHER OUTCOMES:
clinical outcomes via RANO criteria (Response Assessment in Neuro-Oncology Criteria) | 0-24 Months
  describe response rates using Response Assessment in Neuro-Oncology Criteria to interpret MRI (magnetic resonance imaging) scans
Biodistribution via PET (Positron-emission tomography) | 0-43 days
  89Zr-KB004 Positron emission tomography imaging will be used

CONTACTS AND LOCATIONS:
Overall Officials: Hui Gan, Principal Investigator — Austin Health
Locations (2):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No